CLINICAL TRIAL: NCT04871152
Title: Trip-tox Study. Analysis of the Efficacy and Satisfaction of Symptomatic Treatment With Triptans in Patients With Chronic Migraine Undergoing onabotulinumtoxinA Treatment
Brief Title: Trip-Tox, Effectiveness of Triptans Before and After Onabotulinumtoxin A Treatment in Chronic Migraine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-TOX-2020-67
Record Dates: First submitted 2021-04-23; First posted 2021-05-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Chronic Migraine
MeSH Terms: interventions — Botulinum Toxins, Type A; Tryptamines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic migraine: In the same group of patients, the response to triptans will be analyzed at 3 different times with respect to the start of treatment with onabotulinumtoxinA: before treatment, after 4 months and after 7 months of treatment.
  Interventions: Drug: OnabotulinumtoxinA

INTERVENTIONS:
Drug: OnabotulinumtoxinA — To compare the effectiveness of triptans before and after initiation of treatment with OnabotuliumtoxinA.
  Other Names: Triptans

SUMMARY:
Observational, longitudinal, prospective, prospective, comparative study of the effectiveness of triptans before and after onabotulintoxin A initiation in a single group of chronic migraine patients.

DETAILED DESCRIPTION:
Hypothesis In patients with chronic migraine the efficacy of triptans, previously taken by the patient for the migraine attack, is better and more satisfactory after starting treatment with onabotulinumtoxinA.

Objectives To analyze the efficacy and satisfaction of the triptan usually taken by the patient with chronic migraine before starting preventive treatment with onabotulinumtoxinA, at 4 months, after two sessions of Botox, and at 7 months of treatment, after three sessions of Botox.

Sample size n=100 patients with chronic migraine in whom treatment with onabotulinumtoxinA is indicated. The indication for Botox treatment will be performed as usual and the patient will take his usual triptan if he has a migraine attack, so there is no therapeutic modification in this study that could involve any bioethical issue.

All patients signed the informed consent and the study was approved by the Comitè d'Ètica de la Investigació amb Medicaments (CEIm) de l'Hospital de la Santa Creu i Sant Pau.

ELIGIBILITY:
Inclusion Criteria:

* ICHD-3 criteria for chronic migraine (code 1.3). See Table 3.
* Older than 18 years and younger than 65 years.
* Migraine started in their lifetime before the age of 50 years.
* Migraine of more than one year of evolution since diagnosis.
* Normal cranial CT/MRI study.
* Indication for treatment with Botox
* Taking triptans as a rescue treatment for migraine attacks

Exclusion Criteria:

* Pregnant women
* Migraine of less than one year of evolution since diagnosis.
* Pathologies that contraindicate the use of OnabotulinumtoxinA (myasthenia gravis, myopathies).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet criteria for chronic migraine and have failed 2 or more oral preventive treatments (including topiramate) or have a contraindication to taking topiramate.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-09-25 (Estimated); Study Completion 2022-09-25 (Estimated)

PRIMARY OUTCOMES:
Change efficacy (Pain free at two hours ) | From baseline to 4 months
  Percentage of patients who are completely free of pain after two hours of ingestion of their usual triptan.
Change efficacy (Pain free at two hours ) | From baseline to 7 months
  Percentage of patients who are completely free of pain after two hours of ingestion of their usual triptan.
Satisfaction (Likert scale 1-5) | From baseline to 4 months
  Satisfaction of treatment with triptans before and after treatment with OnabotulinumtoxinA
Satisfaction (Likert scale 1-5) | From baseline to 7 months
  Satisfaction of treatment with triptans before and after treatment with OnabotulinumtoxinA

SECONDARY OUTCOMES:
Pain free at one hour | 4 and 7 months
  Percentage of patients who are completely free of pain after one hour of ingestion of their usual triptan.
Sustained pain-free | 4 and 7 months
  Percentage of patients who achieve pain-free at two hours and do not require rescue medication within 24-48 hours.
Headache relapse | 4 and 7 months
  Percentage of patients experiencing recurrence of pain within 48 h on triptans with long half-life or 24 h on triptans with short half-life.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Belvís, PhD, Principal Investigator — Fundació de Gestió Sanitària de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Headache and Neuralgia Unit. Neurology Department. Hospital Santa Creu i Sant Pau, Barcelona, Spain